CLINICAL TRIAL: NCT05061875
Title: Pharmacokinetics of Ceftriaxone Free Fraction Administered at High for the Treatment of Serious Infections
Brief Title: Pharmacokinetics of Ceftriaxone Free Fraction
Acronym: Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-CEF-2021-01
Record Dates: First submitted 2021-09-13; First posted 2021-09-30 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-02

CONDITIONS: Ceftriaxone Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients treated with ceftriaxone doses equal to or higher 4 grams / day.

SUMMARY:
Prospective observational follow-up study for the study and modeling of the pharmacokinetics of the free fraction of ceftriaxone in patients treated with high doses of ceftriaxone (greater than or equal to 4 grams per day).

DETAILED DESCRIPTION:
A prospective follow-up observational study to study and model the pharmacokinetics of the ceftriaxone free fraction in patients treated with high doses of ceftriaxone (greater than or equal to 4 grams per day). it is a pilot study that has between 10 and 20 patients. This study will not condition the treatment of patients at any time.

The samples will be processed after their extraction. The concentration of the samples will be analyzed using a high-performance gilent infinity liquid chromatograph coupled to a mass spectrometer using positive or negative ionization using electrospray.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 55 years of age receiving treatment with high-dose ceftriaxone (minimum 4 grams / day) for any clinical indication in the study period.
* Creatinine <1.5 mg / dL
* The patient must have received at least 48 hours of treatment with the same previous therapeutic regimen to extraction.
* The subject or her representative must give their verbal or written consent to participate in the study. East Consent can be revoked at any time without prejudice to the patient.

The consent it will be recorded in your medical record.

Exclusion Criteria:

* Patients under 55 years of age.
* Creatinine> 1.5 mg / dL
* Patient with less than 48 hours of treatment with high-dose ceftriaxone.
* Subjects with allergy or hypersensitivity to cephalosporins and penicillins.
* Subjects who do not grant or withdraw their consent.
* Patients whose concomitant treatment presents possible interactions with the study medication. The possible interactions will be evaluated by staff of the Pharmacy Service.

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with ceftriaxone doses equal to or higher 4 grams / day. This study will in no case condition the treatment of patients.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration [Cmax] | Up to 24 weeks.
  Determine the maximum plasma concentration of ceftriaxone after the administration of high doses (equal to or greater than 4 grams / day).

SECONDARY OUTCOMES:
To determine the plasma concentration of the free fraction of ceftriaxone 24 hours after the administration of the daily dose (trough level) in patients receiving doses equal to or greater than 4 grams / day. | Up to 24 weeks.
  Plasma concentration of the free fraction of ceftriaxone after 24 hours of the start of the daily dose (trough level) in patients treated with doses at or above 4 grams / day.
Determine the plasma concentration of the free fraction of ceftriaxone during 24 hours in patients receiving doses equal to or greater than 4 grams / day. | Up to 24 weeks.
  Plasma concentration of the free fraction of ceftriaxone for 24 hours in patients receiving doses equal to or greater than 4 grams / day.
Ceftriaxone plasma clearance. | Up to 24 weeks.
  determine the plasma clearance of ceftriaxone in patients receiving doses equal to or greater than 4 grams / day.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Victoria Gil Navarro, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain